CLINICAL TRIAL: NCT01256151
Title: Open-label, Randomized, Single-Dose, 2 Way Crossover Bioequivalence Study Comparing A New Alprazolam Sublingual Tablet Formulation To A Reference Alprazolam Immediate Release Tablet
Brief Title: Pharmacokinetics Of Alprazolam Sublingual Tablet Versus Conventional Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A6131024
Record Dates: First submitted 2010-12-06; First posted 2010-12-08 (Estimated); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Anxiety Disorder
Keywords: Bioequivalence; sublingual; alprazolam; pharmacokinetics
MeSH Terms: conditions — Anxiety Disorders | interventions — Alprazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alprazolam conventional tablet (Active Comparator): Alprazolam conventional tablet
  Interventions: Drug: Alprazolam tablet
- Alprazolam sublingual tablet (Experimental): Alprazolam sublingual tablet
  Interventions: Drug: Alprazolam sublingual

INTERVENTIONS:
Drug: Alprazolam tablet — 1 mg single dose of alprazolam conventional tablet
  Arms: Alprazolam conventional tablet
Drug: Alprazolam sublingual — 1 mg single dose of alprazolam sublingual tablet
  Arms: Alprazolam sublingual tablet

SUMMARY:
To assess if the sublingual tablet will have similar pharmacokinetics as the conventional tablet of alprazolam.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2.
* Signed informed consent.

Exclusion Criteria:

* Evidence or history of clinically significant abnormalities
* Positive drug screen, excessive alcohol and tobacco use

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) from time zero to last measurable time of alprazolam | 72 hours
Peak concentration of alprazolam | 72 hours

SECONDARY OUTCOMES:
Area under the curve from time zero to infinity | 72 hours
AUC% extrapolated | 72 hours
Time of Cmax | 72 hours
half-life of alprazolam | 72 hours
Clinically significant safety laboratory tests | Screening, Day 0, Day 4
Clincally significant vital signs | Screening, Day 4
Clinically significant adverse events | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New Haven, Connecticut, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6131024&StudyName=Pharmacokinetics%20Of%20Alprazolam%20Sublingual%20Tablet%20Versus%20Conventional%20Tablet